CLINICAL TRIAL: NCT01853280
Title: L-methylfolate Supplementation to OROS-Methylphenidate Pharmacotherapy in ADHD Adults: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial
Brief Title: L-methylfolate Supplementation to OROS-Methylphenidate Pharmacotherapy in ADHD Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pamlab, Inc. (Industry)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-P-000379
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; Deplin; L-methylfolate; Natural Treatments; Medical Food
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 5-methyltetrahydrofolate; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Methylfolate (Experimental): 15 mg of L-Methylfolate (Deplin®) daily for 12 weeks as a supplement to OROS-Methylphenidate.
  Interventions: Drug: L-methylfolate; Drug: OROS-Methylphenidate
- Placebo (Placebo Comparator): 15 mg matched placebo comparator, with open-label OROS-Methylphenidate
  Interventions: Drug: OROS-Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: L-methylfolate — 15mg/day L-methylfolate.
  Other Names: Deplin®
  Arms: L-Methylfolate
Drug: OROS-Methylphenidate — All subjects will be treated with open-label OROS-MPH
  Other Names: Concerta®
Drug: Placebo — 15 mg matched placebo comparator, with open-label OROS-Methylphenidate
  Arms: Placebo

SUMMARY:
This pilot study seeks to evaluate initial evidence for the effect of L-methylfolate supplementation to OROS-Methylphenidate pharmacotherapy on ADHD symptoms and associated features in adults with ADHD, as well as tolerability of this supplementation. The investigators will conduct a 12-week double-blind randomized placebo-controlled trial with L-methylfolate supplementing open-label OROS-Methylphenidate (OROS-MPH). The investigators propose to examine 40 adult (ages 18-55) subjects satisfying the DSM-IV diagnostic criteria for ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ages 18-55 years of age.
2. A diagnosis of childhood onset ADHD, meeting all but the age of onset criteria according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), based on clinical assessment. Childhood onset will be defined according to established research criteria, requiring onset of two symptoms of inattentive or of impulsive/hyperactive traits by the age of 12.
3. A score of 24 or more on the Adult ADHD Investigator Symptom Report Scale (AISRS).

Exclusion Criteria:

1. A history of non-response or intolerance to methylphenidate at adequate doses as determined by the clinician.
2. A history of intolerance to L-methylfolate supplementation.
3. Pregnant or nursing females.
4. Serious, unstable medical illness including hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrinologic (thyroid), neurologic (seizure), immunologic, or hematologic disease.
5. Glaucoma.
6. Clinically unstable psychiatric conditions including suicidality, homicidality, bipolar disorder, psychosis, history of or current marked anxiety, tension or agitation potentially exacerbated by a stimulant, or lifetime history of any other clinically serious condition potentially exacerbated by a stimulant, such as mania or psychosis.
7. Significant impairment due to tics, based on clinician judgment.
8. A family history or diagnosis of Tourette's syndrome
9. Current (within 3 months) DSM-IV criteria for abuse or dependence with any psychoactive substance other than nicotine.
10. Multiple adverse drug reactions.
11. Any other concomitant medication considered to be effective for management of ADHD; individuals on stable treatment with agents with central nervous system activity will be allowed to participate, as detailed in the Concomitant Medication portion of the protocol.
12. Current use of MAO Inhibitor or use within the past two weeks.
13. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
14. Use of supplemental folic acid greater than 400 mcg per day, L-methylfolate, or Omega-3 Fatty Acids greater than 800 mg per day within two weeks prior to the baseline study visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total enrollment number (those who signed informed consent) was 47, however, 3 subjects were either found ineligible or lost to follow up before they could be assigned to an arm of the study. Thus 44 subjects were randomized to the study.
Groups:
- L-Methylfolate: 15 mg of L-Methylfolate (Deplin) daily for 12 weeks as a supplement to OROS-Methylphenidate.
- Placebo (for L-Methylfolate): 15 mg matched placebo comparator with open-label OROS-Methylphenidate
Period: Overall Study
Arm/Group | L-Methylfolate | Placebo (for L-Methylfolate)
Started | 22 | 22
Completed | 20 | 16
Not Completed | 2 | 6
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-Methylfolate | Placebo (for L-Methylfolate) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.4) | 37.7 (8.9) | 39.96 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 17 | 36
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: The AISRS is an 18-item questionnaire administered by the clinician assessing each of the individual DSM-IV symptoms of ADHD. Each symptom is rated on a scale of severity from 0 (none) to 3 (severe), and the 18 symptom questions are summed to calculate a total score. The minimum total score is a 0, while the maximum total score is a 54. The AISRS was compared from baseline to completion, over the course of the 12 week study.
Time Frame: 12 weeks
Population: While 44 subjects were randomized to receive the study drug, only 41 subjects actually began taking the medication, and as such were evaluated using the AISRS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-Methylfolate | Placebo (for L-Methylfolate)
Number analyzed (Participants) | 22 | 19
units on a scale | -22.9 (10.4) | -20.8 (11.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the entire time subjects were enrolled in the study beginning as their screening visit and ending at their week 12 completion visit.
Arm/Group | L-Methylfolate | Placebo (for L-Methylfolate)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 20/22 | 19/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Methylfolate (N=22) | Placebo (for L-Methylfolate) (N=22)
Headache (Nervous system disorders) | 17 (40) | 6 (12)
Insomnia (Nervous system disorders) | 11 (24) | 8 (16)
Sedation (Nervous system disorders) | 3 (3) | 3 (3)
Cold/Infection/Allergy (Infections and infestations) | 12 (17) | 6 (11)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (19) | 7 (8)
Decreased Appetite (Gastrointestinal disorders) | 7 (15) | 10 (29)
Tense/Jittery (Nervous system disorders) | 6 (11) | 3 (3)
Nausea/Vomit/Diarrhea (Gastrointestinal disorders) | 6 (18) | 7 (10)
Neurological (Nervous system disorders) | 1 (1) | 3 (5)
Decreased energy (General disorders) | 1 (1) | 0 (0)
Mucosal Dryness (Nervous system disorders) | 6 (15) | 10 (25)
Anxious/worried (Psychiatric disorders) | 4 (6) | 3 (5)
Agitated/irritable (Psychiatric disorders) | 1 (4) | 4 (5)
Sad/down (Psychiatric disorders) | 3 (5) | 5 (5)
Cardiovascular (Cardiac disorders) | 3 (3) | 3 (11)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Genitourinary (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Dizzy/lightheaded (Nervous system disorders) | 0 (0) | 3 (3)
Autonomic: Drool/sweat (Nervous system disorders) | 0 (0) | 2 (5)
Tics (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT01853280/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT01853280/SAP_001.pdf